CLINICAL TRIAL: NCT02597322
Title: An Open-label, Non-randomized, Multicenter, Two Stage Designed Phase II Study of Axitinib for Downstaging Large Renal Tumors Not Primarily Suitable for Partial Nephrectomy (AXIPAN)
Brief Title: Study of Axitinib for Downstaging Large Renal Tumors Not Primarily Suitable for Partial Nephrectomy (AXIPAN)
Acronym: AXIPAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P110209
Record Dates: First submitted 2015-06-08; First posted 2015-11-05 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2017-03

CONDITIONS: cT2a N0NxM0 Renal Tumor
Keywords: Axitinib; T2a Renal tumor; organ confined tumors; nephron sparing surgery; nephron sparing procedure; radical nephrectomy
MeSH Terms: interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AXITINIB (Experimental)
  Interventions: Drug: AXITINIB

INTERVENTIONS:
Drug: AXITINIB — Axitinib is an oral, potent, and selective inhibitor of vascular endothelial growth factor (VEGF) receptors 1, 2, 3 It will be supplied as 1 mg and 5 mg film coated tablets for oral administration in light protecting bottles of 60 tablets.
  Other Names: AG013736

SUMMARY:
Axitinib (AXITINIB) is an oral, potent, and selective inhibitor of vascular endothelial growth factor receptors 1, 2, and 3 which has achieved objective response rate of 44.2% in phase II study in cytokine-refractory metastatic renal-cell cancer patients.

Pre-surgical treatment with Axitinib could allow a substantial proportion of patients with large organ confined tumors to benefit from NSS.

The Objective is to determine the efficacy of Axitinib administered prior to surgery in patients with large organ confined tumors not primarily suitable for NSS (cT2aNoNxM0) for shifting from a radical nephrectomy indication to a nephron sparing procedure.

DETAILED DESCRIPTION:
Radical nephrectomy (RN) is the current standard of care for large organ confined renal tumors.

Experience and surgical technical improvements have allowed the feasibility of Nephron Sparing Surgery (NSS) in tumors larger than 4 cm and up to 7cm. Very limited data exist regarding the feasibility and safety of NSS in tumors larger than 7cm.

It has been demonstrated that NSS compared to RN offers similar oncological outcome while better preserving renal function and thus improving overall survival.

The purpose of this study is to test the possibility of offering patients with large organ confined renal tumors, candidates for radical nephrectomy according to current guidelines the benefit of partial nephrectomy thanks to axitinib neo-adjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must sign IRB/EC-approved informed consent.
* Age ≥ 18
* Histologically proven clear cell RCC (obtained by CT or US guided biopsy)
* cT2a N0NxM0 Renal tumor according to 2009 TNM classification (tumor Ø> 7cm; ≤ 10 cm)
* No evidence of preexisting uncontrolled hypertension as documented by 2 baseline blood pressure readings taken at least 1 hour apart.
* Normal renal function (MDRD creatinin clearance ≥ 60 ml/min)
* Patients must have adequate organ function defined as: Platelets ≥ 150 x 109/L, hemoglobin > 9 g/dl, absolute neutrophil count (ANC) >1.5 x 109/L; Bilirubin < 2 mg/dL, aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 times the upper limit of normal; Total cholesterol ≤ 9.1 mmol/l and triglyceride level ≤ 4.5 mmol/l
* Urinary protein <2+ by urine dipstick.
* Patients with reproductive potential must use medically acceptable contraceptive method.
* Beneficiary of a social coverage (except AME)

Exclusion Criteria:

* Patients with < 50 % clear cell histology
* Evidence of locally advanced disease: cT stage≥T2b, N Stage≥1 or metastatic disease (M1)
* Patients must not be pregnant or lactating.
* Patients must not have uncompensated coronary artery disease or an history of myocardial infarction or severe or unstable angina within the past six months or severe diabetes mellitus with severe arterial peripheral disease or deep venous or arterial thrombosis or embolism with the past 3 months. Patients must not need curative anticoagulants.
* Patients must not have any medical/systemic or psychiatric disorder incompatible with the study.
* Patients must not have a history of significant gastric or small bowel resection, malabsorption syndrome, or other lack of integrity of the upper gastrointestinal tract that may compromise the absorption of Axitinib or an unavailability of the oral route.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-02; Primary Completion 2015-11 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The number of patients actually experiencing a partial nephrectomy for a tumor ≤ 7cm | At 6 months after beginning of the treatment

SECONDARY OUTCOMES:
Response rate according to RECIST criteria | At 30 months after beginning of the treatment
Number of participants with treatment-related serious adverse events and their grades according to CTCAE V4.0. | At 30 months after beginning of the treatment
Renal function assessed by serum creatinin | At baseline and at 30 months after beginning of the treatment
Renal function assessed by calculated glomerular filtration rate (GFR) according to MDRD formula | At baseline and at 30 months after beginning of the treatment
Renal function assessed by renal scintigraphy | At baseline and at 30 months after beginning of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean Jacques Patard, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris, Bicêtre Hospital
Locations (1):
- Bicêtre Hospital, Le Kremlin-Bicêtre, France